CLINICAL TRIAL: NCT03710213
Title: Automated Text Message Navigation to Improve Outpatient Colonoscopy Show Rate and Bowel Preparation
Brief Title: Automated Navigation to Improve Outpatient Colonoscopy Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Shivan J Mehta, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 831701
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Adherence, Patient; Colonoscopy; Text Messaging
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care includes (1) bowel preparation instructions that are delivered via mail or through a secure online messaging portal, (2) a phone call from the endoscopy staff in the week prior to colonoscopy, and (3) the option to call the endoscopy staff during business hours to have any questions answered on demand.
- Text Message-based Intervention (Experimental): In addition to usual care, the text message-based intervention consists of the subject receiving text messages per a pre-determined protocol starting 7 days prior to the date of scheduled colonoscopy, in addition to two text messages at the time of enrollment explaining the texting program. Of note, if a patient in the intervention arm cancels or reschedules their colonoscopy after randomization, they will not receive any additional protocol text messages as part of this trial.
  Interventions: Behavioral: Text Message-based Intervention

INTERVENTIONS:
Behavioral: Text Message-based Intervention — The intervention consists of a series of educational and reminder text messages that a patient will receive in the week prior to a scheduled colonoscopy, in addition to two text messages at the time of enrollment explaining the texting program.
  Arms: Text Message-based Intervention

SUMMARY:
Outpatient colonoscopy adherence is negatively impacted by poor communication and challenges with bowel preparation. We plan to perform a randomized controlled trial at the Pennsylvania Presbyterian Medical Center to (1) provide text message-based educational and reminder messages to patients regarding a scheduled colonoscopy, and (2) evaluate the impact of the texting intervention on colonoscopy show rate and bowel preparation.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of cancer death in the US, yet there are effective screening and treatment strategies that allow for early detection and treatment. CRC screening is recommended for all individuals aged 50-75, which could include stool testing or colonoscopy, but national rates are still suboptimal at 59-65%. Colonoscopy is an essential component of CRC screening, as it is also required if stool testing is positive. However, colonoscopy requires a complex process to identify an escort, purchase the preparation, take a day off from work, adhere to a clear liquid diet, and complete the split-dose preparation as recommended. This results in a significant no-show and cancellation rate, along with suboptimal preparation quality, which can lead to non-adherence and incomplete screening.

Current approaches to engaging patients include having nurses call patients before the procedure or patient navigators. However, it is often difficult to get patients on the phone, and these interventions can be costly, making it less scalable for clinical practices. Other interventions such as videos or mobile apps have been limited by poor user experience or limited engagement with the patient. There is an opportunity to leverage an automated text message navigation intervention using the Way to Health (WTH) platform to improve patient engagement prior to colonoscopy completion. The WTH platform is a Penn Medicine platform that is hosted on site at the University of Pennsylvania. The platform allows custom text messages to automatically be sent to patients, in addition to bidirectional message capabilities. WTH is protected by a secure firewall and is a HIPAA compliant platform.

In the past year, our team conducted a quality improvement pilot initiative using WTH that tested the feasibility and impact of a one-week text messaging protocol for patients who were scheduled for outpatient colonoscopy. The text messages sent to patients contained information about the preparation process and instructions, expectations about the procedure, and reminders about location and timing. Among the 21 patients enrolled in the pilot, we found high user acceptability and higher colonoscopy show rates as compared to baseline values at Pennsylvania Presbyterian Medical Center. As such we believe that the texting intervention is feasible for testing in the context of a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for outpatient colonoscopy at Pennsylvania Presbyterian Medical Center
* Subject has a cell phone with enabled text messaging capability

Exclusion Criteria:

* Fewer than 14 days between the time of enrollment and time of scheduled colonoscopy
* Subject is non-English speaking requiring a translator
* Subject is not the primary individual receiving the text messages

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Colonoscopy show rate with good or excellent bowel prep | Assessed on day of colonoscopy
  The proportion of patients who show up to their scheduled colonoscopy appointment and have a good or excellent prep

SECONDARY OUTCOMES:
Colonoscopy show rate | Assessed on day of colonoscopy
  The proportion of patients who show up to their scheduled colonoscopy appointment
Bowel preparation quality | Assessed on day of originally-scheduled colonoscopy
  The grading of bowel preparation quality (poor, fair, adequate, good, excellent) among those patients who show to their scheduled colonoscopy
Colonoscopy cancellation rate | Assessed on day of originally-scheduled colonoscopy
  The proportion of patients who cancel their originally scheduled colonoscopy appointment
Colonoscopy reschedule rate | Assessed on day of originally-scheduled colonoscopy
  The proportion of patients who cancel and reschedule (for a future date) on the same day, at least one day prior to the originally scheduled colonoscopy appointment date
Colonoscopy no-show rate | Assessed on day of originally-scheduled colonoscopy
  The proportion of patients who do not show for their scheduled colonoscopy appointment and who have not canceled
Timing of advance cancellation notification (in days) | Assessed on day of originally-scheduled colonoscopy
  The number of days in advance that a patient cancels their scheduled colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Hospital System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahmud N, Asch DA, Sung J, Reitz C, Coniglio MS, McDonald C, Bernard D, Mehta SJ. Effect of Text Messaging on Bowel Preparation and Appointment Attendance for Outpatient Colonoscopy: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jan 4;4(1):e2034553. doi: 10.1001/jamanetworkopen.2020.34553. PMID 33492374

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT03710213/Prot_SAP_000.pdf